CLINICAL TRIAL: NCT07396012
Title: Relation Between Degree of Lumbar Spine Curvature and Dynamic Knee Valgus in Smartphone Addict With Non-specific Low Back Pain
Brief Title: Relation Between Degree of Lumbar Spine Curvature and Dynamic Knee Valgus in Smartphone Addicts
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dawlat Mazen Mahmoud Zidan, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/006139
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smartphone Addict With Non Specific Low Back Pain: Sixty-eight subjects who are Smartphone Addict With Non Specific Low Back Pain and aged from 18 to 25 years old will be allocated into one group

INTERVENTIONS:
Other:

SUMMARY:
The purpose of this study will be to investigate the relation between degree of lumbar spine curvature and dynamic knee valgus angle in smartphone addict students with non-specific low back pain.

DETAILED DESCRIPTION:
Smartphone usage can potentially cause musculoskeletal disorders in the lower back. Continuous smartphone use has been shown to create proprioception impairments in the cervical vertebra and postural alterations in the cervical and lumbar vertebrae (slouched posture)

Understanding the relationship between lumbar spine curvature (hyperlordosis, hypolordosis) and knee valgus angle is crucial for:

1. Preventing Musculoskeletal Disorders

   * Excessive knee valgus increases knee injury risk.
   * Abnormal lumbar curvature (hyper lordosis) may alter lower limb kinematics, contributing to knee malalignment.
2. Improving Rehabilitation Strategies: If lumbar posture influences knee mechanics, interventions (such as core stabilization) could reduce valgus and injury risk.
3. Ergonomics: Sedentary lifestyles and poor posture may exacerbate both spinal misalignment and knee valgus, increasing osteoarthritis risk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from both genders with an age range between 18 and 25 years old.
* Sound physical and mental health.
* Body mass index 18.5 to 24.9 kg/m2.
* Subjects with chronic low back pain. Smart phone addiction.

Exclusion Criteria:

* Stroke
* Balance problems
* Visual problems
* Any other physical disorder that may affect our measurement
* Pregnancy
* Obesity
* Comorbidities such as cardiovascular or respiratory conditions

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty-eight subjects who are smart phone addicted with non specific low back pain and are aged from 18 to 25 years old will be allocated into one group.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Lumbar spinal curvature | 8 weeks
  Kinovea software program will be used to assess lumbar curvature mainly the cobb angle of lumbar lordosis.
  Colored markers can be placed on key anatomical landmarks ( spinous processes of L1-L5) while the subject stands in a relaxed, natural posture with feet shoulder-width apart.
  the image will be captured from a lateral (side) view of the spine. and the Kinovea software will analyze and measure angle. Normal Lumbar Lordosis: ~30-60° (varies by method), hyperlordosis: >60° (excessive curvature), hypolordosis (Flat Back): <30° (reduced curvature).

SECONDARY OUTCOMES:
Assessment of pain intensity | 8 weeks
  A visual analogue scale (VAS) will be used to measure the intensity of low back pain. With a score of 0 for no pain and 10 for the worst pain ever. Patients rated their level of pain as mild if they scored 3.4 or less, moderate if they scored 3.5 to 7.4, and severe if they scored 7.5 or higher.
Assessment of smart phone addiction | 8 weeks
  The smart phone addiction scale (SAS) will be used to assess smartphone addiction.
  This is a valid and reliable 10-question measure for diagnosing smartphone addiction. Each question has a potential value ranging from 1 to 6, and the overall questionnaire score can range from 10 to 60 points. A score of 34 is regarded a cut-off for smartphone addiction, with higher values suggesting stronger addiction.
Assessment of quadriceps muscle strength | 8 weeks
  Hand held dynamometer will be used to assess quadriceps muscle strength. The patient sat on a chair with 90° hip/knee flexion; dynamometer placed 2-5 centimeters above malleoli on anterior tibia. the patient will be asked to push your leg forward as hard as possible.
  Test execution:
  Contraction Type: Isometric (hold 3-5 seconds (sec)). Trials: 3 repetitions (30-sec rest between trials). Recording: Peak force from the best of 3 trials. Normal measuring: Men: ~35-45 kg (77-99 lbs). Women: ~25-35 kg (55-77 lbs)
Assessment of dynamic knee valgus angle | 8 weeks
  Kinovea software will be used to assess the dynamic knee valgus angle from a frontal view during a single-leg squat. Marks will be placed on hip at anterior superior iliac spine, Knee midpoint, and ankle midpoint. Measure the angle between the hip-knee-ankle line (180° = neutral, <180° = valgus). The depth of the squat task to 60°will be determined by placing a block behind the participant, and the gluteal muscles contact the block at 60° knee flexion. The non-dominant leg will be held with 90° knee flexion and 45° hip flexion during the whole task. The test will be considered successful if: 1) the person maintains the correct position during the test; 2) he performs the test at the predetermined pace; 3) the suspended leg does not touch the ground; 4) the heel of the dominant foot rests on the ground.

CONTACTS AND LOCATIONS:
Overall Officials: Rabab Monged, PHD, Study Director — October 6 University; Alaa Balbaa, Professor, Study Chair — Cairo University
Locations (1):
- Dawlat Mazen Mahmoud, Giza, Egypt